CLINICAL TRIAL: NCT06024876
Title: A Clinical Study Evaluating the Safety and Efficacy of Ex-vivo tBE Edited Autologous Hematopoietic Stem Progenitor Cells (CS-101) in Treating Subjects With β-thalassemia
Brief Title: A Clinical Study Evaluating the Safety and Efficacy of CS-101 in Treating Subjects With β-thalassemia
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: CorrectSequence Therapeutics Co., Ltd (Industry)
Collaborators: First Affiliated Hospital of Guangxi Medical University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CS-101-06
Record Dates: First submitted 2023-08-23; First posted 2023-09-06 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Beta-Thalassemia
MeSH Terms: conditions — beta-Thalassemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CS-101 (Experimental): CS-101: Autologous CD34+ hematopoietic stem cell suspension modified by ex vivo base editing technique
  Interventions: Biological: CS-101

INTERVENTIONS:
Biological: CS-101 — Autologous CD34+ hematopoietic stem cell suspension modified by ex vivo base editing technique

SUMMARY:
The goal of this open label, single-arm clinical study is to learn about the safety and efficacy of CS-101 in treating β-thalassemia.

DETAILED DESCRIPTION:
CS-101 is an autologous CD34+ cell suspension, edited by ex vivo base editing technology, which modifies the BCL11A binding site in HBG promoter, so that it loses the ability to bind to BCL11A, which can re-induce the production of γ-globin chain and increase the concentration of fetal hemoglobin(HbF) in the blood, compensating for the function of missing adult hemoglobin HbA to achieve clinical cure. The therapy addresses two major challenges in the current treatment of the disease: lack of matching donors and graft-versus-host diseases in allogeneic hematopoietic stem cell transplantation.

ELIGIBILITY:
Key Inclusion Criteria：

* 6 to 35 years old(inclusive) male or female subjects at the time of informed consenting
* Diagnosis of β-thalassemia, genotypes include but are not limited to β+β0，βEβ0，β0β0, etc
* History of at least≥8 units/year of packed RBC transfusions in the prior 12 months prior to the screening period
* Generally in good condition, Karnofsky performance score≥60 points for subjects≥16 years old at the time of autologous hematopoietic stem cell collection, or Lansky Play-Performance score≥60 points for subjects under 16 years old, or equivalent clinical evaluation as the investigator site's common practice

Key Exclusion Criteria:

* Treatment with other investigational medications or other experimental interventions 30 days prior to signing informed consent or within 6 half-lives of the drug, whichever is longer.
* Subjects who have received or are receiving thalidomide and/or Luspatercept, when their drug-drug interaction on the efficacy and safety of CS-101 cannot be ruled out, unless at least there are 3 test results showing the total hemoglobin level before transfusion is below 9g/dL in the past 6 months before screening.
* Previously received allogeneic hematopoietic stem cell transplantation or gene(edited) therapy.
* Subjects have available related fully matching donors and are eligible and prepared for allogeneic hematopoietic stem cell transplantation.
* Those with active infections, including but not limited to: HIV, hepatitis B, hepatitis C, cytomegalovirus, Epstein-Barr virus and treponema pallidum test positive, or known tuberculosis, parasitic infection, etc. who are judged by the investigator to be unsuitable to participate in this study.
* Echocardiography results with ejection fraction below 45%.
* Advanced liver disease, defined as：

Aspartate aminotransferase (AST), alanine aminotransferase (ALT) >3 × upper limit of normal (ULN) or:

Baseline International Normalized Ratio (INR) >1.5 × ULN.

* MRI during the screening period showed heavy iron overload and is judged by the investigator to be unable to participate in the study.

Ages: 6 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 5 (Actual)
Dates: Start 2023-08-26 (Actual); Primary Completion 2025-07-01 (Actual); Study Completion 2025-07-01 (Actual)

PRIMARY OUTCOMES:
Frequency and severity of adverse events(AEs）as assessed by CTCAE v5.0 | From signing informed consent to 12 months post-CS-101 infusion
Time to neutrophil and platelet engraftment | Days post-CS-101 infusion
  Time to neutrophil engraftment is defined as first day of 3 consecutive measurements of absolute neutrophil count≥0.5×10^9/L on three different days； Time to platelet engraftment is defined as first day of 3 consecutive measurements of absolute platelet count≥20×10^9/L on three different days and without platelet transfusion in the past 7 days；
Proportion of subjects with engraftment | within 42 days post-CS-101infusion
  Subjects with engraftment is defined as neutrophil engrafted
Incidence of transplant-related mortality | From baseline to 100 days post-CS-101 infusion
All-cause mortality | From signing informed consent to 12 months post-CS-101 infusion
Proportion of subjects achieving transfusion independence for at least 6 consecutive months | From 3 months up to 12 months post-CS-101 infusion
Time to last red blood cell(RBC) transfusion | Days post-CS-101 infusion

SECONDARY OUTCOMES:
Change in total hemoglobin(Hb) concentration over time | up to 12 months post-CS-101 infusion
  Total hemoglobin concentration change from baseline to 12 months post-CS-101 infusion
Change in fetal hemoglobin(HbF) concentration over time | up to 12 months post-CS-101 infusion
  fetal hemoglobin concentration change from baseline to 12 months post-CS-101 infusion
Chimerism level in Peripheral blood and bone marrow | up to 12 months post-CS-101 infusion
  Proportion of alleles with intended genetic modification in peripheral blood leukocytes and bone marrow over time

CONTACTS AND LOCATIONS:
Overall Officials: Yongrong Lai, M.D., Principal Investigator — First Affiliated Hospital of Guangxi Medical University
Locations (1):
- The First Affiliated Hospital of Guangxi Medical University, Nanning, China